CLINICAL TRIAL: NCT02656446
Title: Accuracy of Depth and Landmark Assessment Using Neuraxial Ultrasound Devices
Status: Completed | Type: Observational
Sponsor: Brendan Carvalho (Other)
Responsible Party: Sponsor-Investigator, Brendan Carvalho, Chief of Obstetric Anesthesia, Professor - Department of Anesthesiology, Stanford University
Organization: Stanford University (Other)
Other Study IDs: 35846
Record Dates: First submitted 2016-01-08; First posted 2016-01-15 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pregnancy
Keywords: Neuraxial; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Accuro Handheld Ultrasound — Use of an Accuro Handheld Ultrasound to identify lumbar interspaces, midline, and depth to epidural space
Device: Standard Ultrasound Machine — Use of standard ultrasound as gold standard to identify lumbar interspaces, midline, and depth to epidural space

SUMMARY:
The purpose of this study is to determine if a handheld ultrasound device helps in the placement of labor epidurals by studying the accuracy of the Accuro Handheld Ultrasound device compared to a standard ultrasound machine.

DETAILED DESCRIPTION:
Pregnant women who present to Labor and Delivery for an anticipated vaginal delivery will be identified as potential participants based on inclusion/exclusion criteria and their desire for labor epidural analgesia. Ultrasound evaluations will be conducted in a cohort of 50 parturients who decide they want epidural analgesia in labor. Prior to epidural placement, a hand held ultrasound device will be utilized to identify L2/3, L3/4 and L4/5 interspace. A mark will be made on the patient's back at these levels. The handheld ultrasound device will also estimate the depth to epidural space at each level using its programmed algorithm. A standard ultrasound will then be used to locate the same interspaces, identify midline, and estimate depth to epidural space with caliper calculation. Upon patient request, an epidural will be placed at L3/4 with a loss of resistance to saline technique. The actual depth to loss of resistance during epidural insertion will be determined by measuring the Tuohy with a sterile measuring tape while it is in the skin.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I, II, or III
* age between 18 and 50
* singleton term pregnancy
* requesting epidural analgesia for anticipated vaginal delivery
* all ethnicities

Exclusion Criteria:

* contraindication for epidural analgesia (bleeding diathesis, neuropathy, severe scoliosis, previous spine surgery, local anesthetic allergy)
* inability to adequately understand the consent form

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 parturients who decide they want epidural analgesia in labor
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Depth to Epidural Space | Within 24 Hours of enrollment
  Determine the difference between the Accuro ultrasound epidural space depth estimation and actual Tuohy epidural depth during epidural insertion at L3/4

SECONDARY OUTCOMES:
Midline Identification | Within 24 Hours of enrollment
  The difference between the Accuro Handheld Ultrasound identification of midline and standard ultrasound machine identification of midline
Interspace Identification | Within 24 Hours of enrollment
  The difference between the Accuro Handheld Ultrasound identification of interspace level and standard ultrasound identification of interspace level
Time to Epidural Placement | Within 24 Hours of enrollment
  Specifically time from insertion of the Tuohy into the skin until removal of the Tuohy after epidural catheter threading
Interspace Levels Attempts | Within 24 Hours of enrollment
  Number of interspace levels attempts for epidural placement
Epidural Failure Rate | Within 24 Hours of enrollment
  Need for replacement epidural or change in anesthetic technique

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, MBBCh, FRCA, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] Carvalho B. Failed epidural top-up for cesarean delivery for failure to progress in labor: the case against single-shot spinal anesthesia. Int J Obstet Anesth. 2012 Oct;21(4):357-9. doi: 10.1016/j.ijoa.2011.06.012. Epub 2011 Nov 22. No abstract available. PMID 22112917
- [Background] Shaikh F, Brzezinski J, Alexander S, Arzola C, Carvalho JC, Beyene J, Sung L. Ultrasound imaging for lumbar punctures and epidural catheterisations: systematic review and meta-analysis. BMJ. 2013 Mar 26;346:f1720. doi: 10.1136/bmj.f1720. PMID 23532866
- [Background] Balki M, Lee Y, Halpern S, Carvalho JC. Ultrasound imaging of the lumbar spine in the transverse plane: the correlation between estimated and actual depth to the epidural space in obese parturients. Anesth Analg. 2009 Jun;108(6):1876-81. doi: 10.1213/ane.0b013e3181a323f6. PMID 19448216
- [Background] Tran D, Kamani AA, Lessoway VA, Peterson C, Hor KW, Rohling RN. Preinsertion paramedian ultrasound guidance for epidural anesthesia. Anesth Analg. 2009 Aug;109(2):661-7. doi: 10.1213/ane.0b013e3181a94c75. PMID 19608844
- [Derived] Seligman KM, Weiniger CF, Carvalho B. The Accuracy of a Handheld Ultrasound Device for Neuraxial Depth and Landmark Assessment: A Prospective Cohort Trial. Anesth Analg. 2018 Jun;126(6):1995-1998. doi: 10.1213/ANE.0000000000002407. PMID 28858898